CLINICAL TRIAL: NCT05599295
Title: A Multicenter, Open-Label, Evaluator-Blinded, Randomized Study to Evaluate the Safety and Tolerability of Single-Dose Intravenous Oritavancin for the Treatment of Pediatric Subjects With Acute Bacterial Skin and Skin Structure Infections
Brief Title: Study to Evaluate the Safety of Intravenous Oritavancin for the Treatment of Children With Skin Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melinta Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Organization: Melinta Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML-ORI-201; 2024-516385-10-00 (EU CTIS Number)
Record Dates: First submitted 2022-10-20; First posted 2022-10-31 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Acute Bacterial Skin and Skin Structure Infection
MeSH Terms: interventions — oritavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Orbactiv (Experimental): Orbactiv will be infused at 15 milligrams/kilogram (mg/kg) over 3 hours for all participants and will not exceed a dose of 1200 mg.
  Interventions: Drug: Orbactiv
- Kimyrsa (Experimental): Kimyrsa will be infused at 15 mg/kg over 3 hours for all participants and will not exceed a dose of 1200 mg.
  Interventions: Drug: Kimyrsa

INTERVENTIONS:
Drug: Orbactiv — Solution for IV infusion
  Other Names: Oritavancin
  Arms: Orbactiv
Drug: Kimyrsa — Solution for IV infusion
  Other Names: Oritavancin
  Arms: Kimyrsa

SUMMARY:
This protocol describes a randomized, open-label study to evaluate the safety and tolerability of 2 formulations of single-dose intravenous (IV) oritavancin diphosphate (Orbactiv and Kimyrsa) for the treatment of pediatric participants with acute bacterial skin and skin structure infections (ABSSSIs).

This study involves 2 oritavancin products, Orbactiv and Kimyrsa. Oritavancin is the active drug substance in both Orbactiv and Kimyrsa. This study protocol distinguishes the differences between Orbactiv and Kimyrsa by providing product-specific data, and information and guidance for Investigators. "Oritavancin" is used to describe drug product data and information and guidance that is not specific to Orbactiv or Kimyrsa (that is, applies to both).

The study involves pharmacokinetic sampling and will evaluate clinical outcome assessments. The study was designed to capture adequate data while minimizing the impact to participants and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 3 months to <12 years of age at randomization
2. Diagnosis of at least 1 of the following ABSSSI infections (known or suspected to be caused by a gram-positive pathogen):

   1. Wound infection: that is either traumatic or surgical in origin, defined as an infection characterized by purulent drainage from a wound with surrounding erythema, edema, and/or induration
   2. Cellulitis/erysipelas: a diffuse skin infection characterized by spreading areas of erythema, edema, and/or induration
   3. Major cutaneous abscess: an infection characterized by a collection of pus within the dermis or subcutaneous tissue that is accompanied by surrounding erythema, edema, and/or induration
3. ABSSSI must present with at least 2 of the following signs and symptoms:

   1. Purulent drainage or discharge
   2. Erythema (>1 centimeter beyond edge of wound or abscess)
   3. Fluctuance
   4. Heat or localized warmth
   5. Edema/induration
   6. Pain or tenderness to palpation

   and at least 1 of the following signs of systemic inflammation:
   1. Proximal lymph node swelling and tenderness
   2. Increased temperature (>38.0°C [>100.4°F])
   3. Decreased temperature (<36.0°C [<96.8°F])
   4. Decreased white blood count (WBC) (<4000/cubic millimeter [mm^3]) or increased WBC (>12,000 mm^3)
   5. Bandemia >10%
   6. C-reactive protein >upper limit of normal (ULN)
4. Written informed consent obtained from parent(s) or legal guardian(s), with written or documented verbal assent of the child obtained, when appropriate, before initiation of any assessments conducted solely for study purposes

Exclusion Criteria:

1. Participants who have received more than 72 hours of effective antibacterial drug therapy for treatment of the current episode of ABSSSI
2. Participants who have received a glycopeptide antibiotic (for example, vancomycin, telavancin, teicoplanin) within 24 hours of randomization
3. Participants who have received dalbavancin within 45 days prior to randomization
4. Participants who have been treated with oritavancin within the last 50 days
5. Participants with infection suspected to be associated with a device or implant
6. Participants with septic shock or hemodynamic instability
7. Participants with ABSSSI due to, or associated with any of the following:

   1. Infection suspected or documented to be caused predominantly by gram-negative pathogens (for example, human or animal bite, injury contaminated with fresh or saltwater, external malignant otitis), fungi, or viruses
   2. Wound infection (surgical or traumatic) or abscess with only gram-negative pathogens
   3. Concomitant infection at another site, not including a secondary ABSSSI lesion (for example, septic arthritis, endocarditis, osteomyelitis). Secondary infections due to the same gram-positive bacteria are eligible to be enrolled in this study.
   4. Infected burn
   5. Primary infection superimposed on a pre-existing skin disease with associated inflammatory changes (for example, atopic dermatitis, eczema)
   6. Any evolving necrotizing process (for example, necrotizing fasciitis), gangrene, or infection suspected or proven to be caused by clostridioides species (for example, crepitance on examination of the ABSSSI site and/or surrounding tissue[s], radiographic evidence of subcutaneous gas in proximity to the infection)
   7. Clinically significant viral infection (for example, influenza, Coronavirus Disease 2019) which, in the investigator's judgement, will impact the study clinical outcome assessments (for example, participant is febrile due to the viral infection)
8. Participants currently receiving chronic systemic immunosuppressive therapy
9. Participants with neutropenia, defined as absolute neutrophil count <500 cells/mm^3
10. Participants with severe renal impairment, defined as an estimated glomerular filtration rate <30 milliliters/minute/1.73 meters squared, using the updated bedside Schwartz formula. For participants under 1 year of age, severe renal impairment is defined as serum creatinine ≥2 times the 97.5th percentile creatinine for age, converted to mg/deciliter or a requirement for dialysis. Participants under 1 year of age with renal impairment require consultation with the sponsor's medical monitor before enrollment.
11. Menstruating females with a positive result for the urine or serum human chorionic gonadotropin test administered at screening
12. Females of childbearing potential (and males with female partners of childbearing potential) unwilling to practice abstinence or use highly effective methods of contraception during the entire study period from the time of the first dose and until 50 days after the last dose of protocol-defined study medication. A list of acceptable methods of contraception is listed in the protocol.
13. Participants with a history of infusion-related immunoglobulin E-mediated allergic reaction or hypersensitivity reaction to glycopeptides (for example, vancomycin, telavancin, dalbavancin, oritavancin, teicoplanin) or any of their excipients
14. Participants who are taking heparin (other than heparin flush for line patency) or warfarin, and/or require anticoagulant monitoring (activated partial thromboplastin time, prothrombin time, international normalized ratio)
15. Participants receiving treatment with an investigational medicinal product or investigational device within 3 months before enrollment or during the study
16. Participants whom the investigator considers unlikely to adhere to the protocol, comply with investigational medicinal product (IMP) administration, or complete the clinical study (for example, unlikely to survive 28 days from initiation of IMP)
17. Participants with alanine aminotransferase or aspartate aminotransferase >3* ULN or total bilirubin ≥2* ULN

Ages: 3 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Day 1 through Day 28

SECONDARY OUTCOMES:
All-cause Mortality | Day 28
Number of Participants with a Clinical Response of Cure or Failure | Day 14 and Day 28
Area Under the Curve of Plasma Concentration (AUC) of Oritavancin | Day 1 (up to 168 hours after start of infusion)
Maximal Plasma Concentration (Cmax) of Oritavancin | Day 1 (up to 168 hours after start of infusion)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (2):
  - Tampa General Hospital, Tampa, Florida
  - Nationwide Children's Hospital, Columbus, Ohio
- Bulgaria (6):
  - Multiprofile Hospital for Active Treatment- Sveti Nikolay Chudotvoretz - LOM EOOD, Lom, Montana
  - Multiprofile Hospital For Active Treatment Dr Tota Venkova, Gabrovo
  - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD-66 Peshtersko Shosse blvd, Plovdiv
  - University Multiprofile Hospital For Active Treatment Kanev AD, Rousse
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine N. I. Pirogov EAD, Sofia
  - University Multiprofile Hospital for Active Treatment - Prof. Dr. Stoyan Kirkovich AD, Stara Zagora
- Greece (3):
  - Attikon University General Hospital, Chaïdári, Attica
  - Hippokratio General Hospital of Thessaloniki, Thessaloniki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- Latvia (2):
  - Daugavpils Regional Hospital, Daugavpils, Daugavpils Aprinkis
  - Children's Clinical University Hospital, Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas, Kaunas County
  - Klaipeda Children Hospital, Klaipėda, Klaipėda County
- Portugal (2):
  - Hospital de Cascais, Alcabideche, Lisbon District
  - Centro Hospitalar de Lisboa Ocidental, EPE - Hospital São Francisco Xavier, Lisbon
- Romania (2):
  - Louis Turcanu Emergency Clinical Hospital for Children, Timișoara, Timiș County
  - Brasov Children Clinical Hospital, Brasov
- Spain (4):
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Sant Joan de Deu - PIN, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid